CLINICAL TRIAL: NCT03146182
Title: Biomarker Guided Antibiotic Treatment in Community-Acquired Pneumonia
Acronym: BIO-CAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gertrud Baunbaek Egelund (Other)
Responsible Party: Sponsor-Investigator, Gertrud Baunbaek Egelund, M.D., Nordsjaellands Hospital
Organization: Nordsjaellands Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIO-CAP_NZH; 2015-002501-11 (EudraCT Number)
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Community Acquired Pneumonia
Keywords: C-reactive protein; Procalcitonin; Community-acquired pneumonia; Antibiotic stewardship
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Patients are treated according to current local guidelines on antibiotic treatment for CAP.
- CRP (Experimental): Patients are treated according to the CRP-algorithm. CRP is measured daily. Antibiotic treatment is stopped when CRP reach threshold value.
  Interventions: Behavioral: CRP-algorithm
- PCT (Experimental): Patients are treated according to the PCT-algorithm. PCT is measured daily. Antibiotic treatment is stopped when PCT reach threshold value.
  Interventions: Behavioral: PCT-algorithm

INTERVENTIONS:
Behavioral: CRP-algorithm — a strategy based on CRP guided antibiotic stewardship
  Arms: CRP
Behavioral: PCT-algorithm — a strategy based on PCT guided antibiotic stewardship
  Arms: PCT

SUMMARY:
The purpose of this study is to determine the efficacy of C-reactive protein and procalcitonin based guidelines versus standard of care to reduce duration of antibiotic exposure in patients hospitalized with community acquired pneumonia.

DETAILED DESCRIPTION:
BIO-CAP is a prospective randomized intervention study which aims to evaluate the efficacy of C-reactive protein (CRP) based guidelines and procalcitonin (PCT) based guidelines to reduce duration of antibiotic exposure in adult patients hospitalized with community-acquired pneumonia (CAP) compared to standard-of-care.

Hypothesis: the duration of antibiotic exposure can be reduced when a biomarker algorithm - in addition to standard of care - is used to stop antibiotic treatment.

1) CRP based guidelines can reduce duration of antibiotic exposure equally to procalcitonin based guidelines and 2) Either of these two biomarker algorithms ( CRP or PCT) are superior compared to standard of care.

Sample size. Preconditions: significance level (α) 5 % and power (β) 80 %. Test: unpaired T-test. Mean treatment time 11 days (SD 5) in this population. Relevant detection limit defined at 2 days. The bonferroni correction has been used to correct for the fact that 2 primary analysis will be performed, why α = 0.005/2 = 0.025. Estimated 100 patient in each arm, thus n = 300.

Site monitoring and auditing. The study is monitored by the unit for Good Clinical Practice, Bispebjerg Hospital, Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older admitted to hospital with community acquired pneumonia defined as a new infiltrate on x-ray and at least one of the following; cough, expectoration, dyspnea, fever and pathological lung-auscultation.
* Not admitted to hospital within the last 14 days
* The patients has been prescribed antibiotic treatment for pneumonia
* The patient can comprehend the written and verbal information and has provided written consent.

Exclusion Criteria:

* Patient are unable to give written consent or patient does not understand the Danish language.
* Active pulmonary tuberculosis
* Severe immunosuppression determined by the treating physician (i.e. treatment with highdose corticosteroid for more than 2 weeks, chemotherapy and neutropenia with neutrophils < 0.5x109/l, ongoing treatment with biological drugs, chronic HIV-infection with CD4 cell count < 350 mio./l, immunosuppression after organ transplantation).
* Pregnancy and breastfeeding
* Patients admitted to hospital and treated against their will.
* Terminal ill patients where active treatment is stopped within the first 48 hours of admission.
* Patients who are, from the date of inclusion, prescribed antibiotic treatment for more than 3 days on a different indication than pneumonia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Duration of antibiotic treatment | 30 days from inclusion
  Number of days in antibiotic treatment for pneumonia

SECONDARY OUTCOMES:
30 day mortality | 30 days from inclusion
  Number of patients who die within 30 days.
Relapse | 30 days from inclusion
  Number of patients who are readmitted due to pneumonia or resumed treatment for pneumonia.

CONTACTS AND LOCATIONS:
Overall Officials: Gertrud B Egelund, M.D., Principal Investigator — Department of pulmonary and infectious diseases, Nordsjaellands Hospital
Locations (1):
- Nordsjællands Hospital., Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: Undecided